CLINICAL TRIAL: NCT00808236
Title: Trans-Nasal Cooling With the RhinoChill Device Following Cardiac Arrest: A Pilot Study
Brief Title: Pre-ROSC Intra-Nasal Cooling Effectiveness
Acronym: PRINCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BeneChill, Inc (Industry)
Responsible Party: Becky Inderbitzen/Vice President Clinical Affairs, BeneChill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-CP1012
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Results first posted 2010-07-16 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Pre-hospital; Mild hypothermia; Resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RhinoChill (Experimental): Intra-arrest cooling with the RhinoChill during advanced cardiac life support
  Interventions: Device: RhinoChill
- Control (Other): Advanced cardiac life support, only
  Interventions: Other: Control

INTERVENTIONS:
Device: RhinoChill — Nasal catheters are placed and cooling is begun during the resuscitation attempt
  Other Names: intra-nasal cooling
  Arms: RhinoChill
Other: Control — Advanced cardiac life support according to American Heart Association & European Resuscitation Council 2005 Guidelines
  Arms: Control

SUMMARY:
The purpose of the study was to demonstrate the safety and feasibility of early intranasal cooling prior to return of spontaneous circulation (ROSC) in the emergency medical services (EMS) environment. It was hypothesized that cooling during the resuscitation attempt would increase ROSC and subsequent survival. The study was not powered to demonstrate statistically-significant differences in any outcome parameter, but was intended as an exploratory study only.

DETAILED DESCRIPTION:
Out of hospital cardiac arrest remains a significant cause of death. Mild hypothermia induced after resuscitation from cardiac arrest has been shown to improve neurologically intact survival. Studies in dogs and rodents have demonstrated improved outcomes when cooling is initiated intra-arrest.

The RhinoChill is a non-invasive cooling device through which rapid cooling is achieved via the intranasal delivery of an evaporative coolant into the nasopharynx. Due to its non-invasive and portable nature, the RhinoChill can be used to begin cooling earlier than other cooling devices.

Studies performed using the RhinoChill in a porcine model of cardiac arrest suggest that cooling with the RhinoChill prior to the first defibrillation attempt facilitates resuscitation and improves resuscitation rate and neurologically intact survival.

This study is being performed to assess the feasibility of using the RhinoChill device in the pre-hospital setting to improve resuscitation from cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Collapse was witnessed
* No pulse
* Unresponsive to external stimuli

Exclusion Criteria:

* Have an etiology of cardiac arrest due to trauma, severe bleeding, drug overdose (OD), cerebrovascular accident (CVA), drowning, smoke inhalation, electrocution, hanging
* Already hypothermic
* Head trauma
* Cannot place intra nasal catheters
* Do Not Attempt to Resuscitate (DNAR) orders
* Known or clinically apparent pregnancy
* Have a known coagulopathy (except therapeutically induced)
* Are known to have a need for supplemental oxygen
* Achieve return of spontaneous circulation (ROSC) prior to initiating cooling
* Are reached by emergency medical services (EMS) personnel more than 20 minutes after collapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Barbut, MD, Study Chair — BeneChill, Inc
Locations (15):
- Belgium (6):
  - CHU St Pierre, Brussels
  - Erasme Hospital (Free University of Brussels), Brussels
  - CHU de Tivoli, La Louvière
  - UZ Gasthuisberg Leuven, Leuven
  - CHR de la Citadelle, Liège
  - Helig Hartzieknehuis Roeselare, Roeselare
- Faculty Hospital Královské Vinohrady, Prague, Czechia
- Germany (6):
  - Medizinisches Zentrum Kreis Aachen gGmbH, Aachen
  - Charite Campus Virchow Klinikum, Berlin
  - Albert Ludwigs University Freiburg, Freiburg im Breisgau
  - Georg August-Universität Göttingen, Göttingen
  - Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
- A.O Ospedale San Gerardo di Monza, Monza, Italy
- Stockholm Prehospital Centrum, Stockholm, Sweden

REFERENCES:
- [Background] Tsai MS, Barbut D, Tang W, Wang H, Guan J, Wang T, Sun S, Inderbitzen B, Weil MH. Rapid head cooling initiated coincident with cardiopulmonary resuscitation improves success of defibrillation and post-resuscitation myocardial function in a porcine model of prolonged cardiac arrest. J Am Coll Cardiol. 2008 May 20;51(20):1988-90. doi: 10.1016/j.jacc.2007.12.057. No abstract available. PMID 18482670
- [Derived] Castren M, Nordberg P, Svensson L, Taccone F, Vincent JL, Desruelles D, Eichwede F, Mols P, Schwab T, Vergnion M, Storm C, Pesenti A, Pachl J, Guerisse F, Elste T, Roessler M, Fritz H, Durnez P, Busch HJ, Inderbitzen B, Barbut D. Intra-arrest transnasal evaporative cooling: a randomized, prehospital, multicenter study (PRINCE: Pre-ROSC IntraNasal Cooling Effectiveness). Circulation. 2010 Aug 17;122(7):729-36. doi: 10.1161/CIRCULATIONAHA.109.931691. Epub 2010 Aug 2. PMID 20679548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by emergency medical system advanced life support personnel over an 8-month period (November 2008 through June 2009). Patients appearing to meet the study criteria were randomized during ongoing resuscitation procedures. Patients that survived to hospital admission were followed until death or hospital discharge.
Pre-assignment Details: Due to the emergency nature of the research, patients were often randomized into the study before all exclusion criteria could be ruled out (e.g., "Do Not Attempt to Resuscitate" (DNAR) orders, drug over-dose (OD), cerebrovascular accident (CVA)). Therefore, patients meeting pre-defined exclusion criteria were not included in the outcome measures.
Groups:
- Control: Advanced cardiac life support (ACLS), only. ACLS procedures were performed in accordance with the European Resuscitation Council 2006 Guidelines.
Period: Overall Study
Arm/Group | RhinoChill | Control
Started | 96 | 104
Met Eligibility Criteria | 84 (Pre-defined exclusions: DNAR(4); had pulse(2); CVA(2); Drug OD(2); On home oxygen(1); Unwitnessed(1)) | 101 (Pre-defined exclusions: Terminal(1); Asphyxia(1), In-hospital(1))
Included in Analysis | 83 (Lost to Follow-Up: taken to non-participating hospital (1)) | 99 (Crossed over & withdrawn (1); Lost to Follow-Up: taken to non-participating hospital (1))
Achieved ROSC | 33 | 43
Admitted to Hospital | 30 (Died during transport to hospital(2); DNAR determination was made at hospital(1)) | 42 (Died during transport to hospital(1))
Completed | 14 | 13
Not Completed | 82 | 91
Not completed — Was not resuscitated | 50 | 56
Not completed — Pre-defined exclusion | 13 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Death | 18 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RhinoChill | Control | Total
Number analyzed (Participants) | 96 | 104 | 200
Age Categorical [Number; unit: participants] — Overall number of participants included in analysis was 181: 82 RhinoChill patients and 99 Control patients
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 35 | 44 | 79
    >=65 years | 47 | 55 | 102
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (13.2) | 64.8 (13.5) | 65 (14)
Gender [Number; unit: participants]
  Female | 23 | 22 | 45
  Male | 59 | 77 | 136
Region of Enrollment [Number; unit: participants]
  Czech Republic | 2 | 4 | 6
  Belgium | 46 | 51 | 97
  Germany | 32 | 33 | 65
  Italy | 3 | 6 | 9
  Sweden | 13 | 10 | 23
Bystander CPR [Number; unit: participants] — The is the number of those participants that received bystander rescue cardiopulmonary resuscitation (CPR) efforts prior to the arrival of emergency medical service (EMS) personnel
  participants
    Received bystander CPR | 31 | 45 | 76
    Did not receive bystander CPR | 51 | 54 | 105
Evaluable Participants [Number; unit: participants] — Eligible participants were those included in the analyses. These excluded those particiapnts found not meet all of the inclusion criteria or to have a pre-defined exclsion criteria as well as those lost to follow-up for whom no data was obtained.
  participants
    Did not meet all Inclusion/Exclusion Criteria | 13 | 3 | 16
    No data obtained | 1 | 2 | 3
    Total evaluable | 82 | 99 | 181
First Rhythm [Number; unit: participants] — First rhythm was defined as ventricular fibrillation/non-perfusing ventricular tacchycardia (VF/VT), asystole, or pulseless electrical activity/electro-mechanical dissociation (PEA/EMD)
  participants
    VF/VT | 24 | 32 | 56
    Asystole | 40 | 44 | 84
    PEA/EMD | 18 | 23 | 41
Elapsed time from collapse until: [Median (Inter-Quartile Range); unit: minutes]
  EMS CPR Initiated | 8 [5 to 10] | 8 [5 to 10] | 8 [5 to 10]
  First Defibrillation Shock (VF only) | 12 [8 to 14] | 12 [7 to 16] | 12 [8 to 15]
  Advanced Life Support (ALS) Arrived | 12 [9 to 16] | 11 [8 to 16] | 12 [9 to 16]
  Intravenous (IV) Access Acquired | 16 [14 to 20] | 15 [12 to 20] | 16 [12 to 16]
  Airway Protected | 18 [14 to 22] | 16 [12 to 20] | 17 [13 to 21]
  Randomized | 20 [16 to 25] | 18 [14 to 22] | 19 [15 to 19]
  Cooling Initiated | 23 [18 to 30] | 113 [71 to 200] | 30 [20 to 64]
  ROSC Achieved | 32 [29 to 38] | 30 [22 to 38] | 31 [23 to 38]
  Arrived at Hospital | 59 [51 to 75] | 60 [42 to 70] | 60 [45 to 71]

OUTCOME MEASURES:

1. Primary Outcome: Achieve Return of Spontaneous Circulation (ROSC)
Description: ROSC was defined as the return of an organized rhythm on electrocardiography (ECG) with a palpable pulse that was maintained for at least 20 minutes.
Time Frame: 1-hour after arrest
Population: Only patients meeting all inclusion/exclusion criteria (IC/EC) were included in the analyses. 15 patients were found to not meet all IC/EC after enrollment. 2 more patients were lost to follow-up and 1 patient was crossed over (Control to RhinoChill) and then withdrawn. Informed consent nor data was obtained for any of these patients.
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 83 | 99
participants | 33 | 43

2. Primary Outcome: Survived to Hospital Discharge
Description: The study end-point was hospital discharge. This outcome measure is the patient count for those that were discharged alive from the hospital.
Time Frame: 30 days after arrest
Population: The set of patients excluding those not meeting IC/EC, not lost to follow-up, or not crossed-over/withdrawn. One RhinoChill patient that achieved ROSC was found to be "DNAR" upon hospital arrival and was excluded from analyses thereafter. The final number of analyzed RhinoChill patients was therefore 82.
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 82 | 99
participants | 14 | 13

3. Primary Outcome: Survived Neurologically-Intact
Description: The Cerebral Performance Categories (CPC) are used to describe neurological outcome. A CPC of 1 or 2 is considered "neurologically intact."
  1. - Good cerebral performance: little to no deficit.
  2. - Moderate cerebral disability: capable of independent activities of daily life
  3. - Severe cerebral disability: conscious, but dependent on others for daily support
  4. - Coma or vegetative state
  5. - Death or brain death
Time Frame: 30-days after arrest
Population: The set of patients excluding those not meeting IC/EC, not lost to follow-up, or not crossed-over/withdrawn.
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 82 | 99
participants | 11 | 9

4. Secondary Outcome: Primary Outcomes in Sub-group With VF/VT as First Rhythm
Description: ROSC, survival, and neurologically-intact survival
Time Frame: hospital discharge
Population: Subset of all included patients with VF/VT as the first cardiac rhythm present upon ECG assessment by EMS personnel
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 24 | 32
participants
  Achieved ROSC | 17 | 21
  Survived to Hospital Discharge | 10 | 10
  Survived Neurologically-Intact | 8 | 6

5. Secondary Outcome: Time to Therapeutic Temperature
Description: The therapeutic temperature range for treatment in cardiac arrest is considered to be 32-34C. Time to therapeutic temperature was taken as the first time in which 34C was measured. Tympanic and core temperatures were taken in all patients.
Time Frame: within 8 hours after enrollment
Population: The subset of patients that were resuscitated and subsequently received in-hospital cooling and reached the designated therapuetic temperatures.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 24 | 32
minutes
  Time to 34C Tympanic Temperature | 102 [81 to 155] | 291 [183 to 416]
  Time to 34C Core Temperature | 155 [124 to 315] | 284 [172 to 471]
  Time to 33C Tympanic Temperature | 170 [101 to 335] | 377 [258 to 635]
  Time to 33C Core Temperature | 315 [180 to 477] | 389 [280 to 649]

6. Secondary Outcome: Length of Stay
Description: Length of stay data for patients admitted to the hospital will be calculated for:
  1. Days on ventilator
  2. Days in intensive care without ventilator
  3. Days in general ward
Time Frame: Hospital Discharge
Population: Evaluable patients admitted to the hospital
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 30 | 42
days
  Non-survivors | 3.0 [2.3 to 5.4] | 2.6 [0.3 to 5.1]
  Survivors - ventilator days | 4.2 [3.0 to 5.8] | 8.8 [5.2 to 11.0]
  Survivors - ICU days (no ventilator) | 2.0 [0.6 to 6.5] | 3.0 [2.0 to 5.0]
  Survivors - general ward days | 12.8 [7.0 to 20] | 11.5 [7.0 to 16]

7. Post Hoc Outcome: Primary Outcomes in Sub-group Receiving EMS CPR Within 10 Minutes of Collapse
Description: ROSC, Survival, and neurologically-intact survival
Time Frame: Hospital discharge
Population: Subset of patients receiving EMS CPR within 10 minutes of collapse (representing 75% of all patients)
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 63 | 74
participants
  Achieved ROSC | 26 | 35
  Survived to Hospital Discharge | 13 | 10
  Survived Neurologically-Intact | 10 | 6

8. Secondary Outcome: Serious Adverse Events (SAEs)
Description: These were defined serious adverse events that are not direct sequelae of the cardiac arrest itself or the underlying cardiac disease. Therefore, these do not include recurrent arrests occcuring within 24 hours of resuscitation nor deaths due to lack of cardiac and/or neurological recovery.
Time Frame: 7 days after arrest
Population: All enrolled patients; see additional modified "at risk" population based on study attrition in the Adverse Event section.
Measure: Number; unit: all participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 96 | 104
all participants | 6 | 12

9. Secondary Outcome: 24-hour Adverse Events (AE)
Description: These were all non-serious adverse events that occurred between the time of enrollment and 24 hours after resuscitation. These did not include a failure to achieve ROSC.
Time Frame: 24 hours after arrest
Population: all enrolled participants
Measure: Number; unit: all participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 96 | 104
all participants
  RhinoChill-related | 17 | 0
  Other | 0 | 3

10. Post Hoc Outcome: Outcomes for Patients Admitted to the Hospital
Description: Suvival and neurologically intact survival
Time Frame: Hospital discharge
Population: Subset of patients that achieved ROSC and were subsequently admitted to the hospital.
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 30 | 42
participants
  Survived to Hospital Discharge | 14 | 13
  Survived Neurologically-Intact | 11 | 9

11. Post Hoc Outcome: Outcomes for VF Patients Admitted to the Hospital
Description: Survival and neurologically-intact survival for patients found in VF/VT admitted to the hospital
Time Frame: Hospital discharge
Population: Subset of patients with an initial rhythm of VF/VT, achieved ROSC and were subsequently admitted to the hospital
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 16 | 21
participants
  All Survivors | 10 | 10
  Neurologically-Intact Survivors | 8 | 6

12. Post Hoc Outcome: Outcomes for Patients Receiving EMS CPR Within 10 Minutes of Collapse That Were Admitted to the Hospital
Time Frame: Hospital Discharge
Population: Subset of patients that received EMS CPR within 10 minutes of collapse, achieved ROSC, and were subsequently admitted to the hospital.
Measure: Number; unit: participants
Arm/Group | RhinoChill | Control
Number analyzed (Participants) | 22 | 34
participants
  Survived to Hospital Discharge | 13 | 10
  Survived Neurologically-Intact | 10 | 6

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected over the first seven days after study enrollment. Other clinically significant adverse events were collected over the first 24 hours.
Description: Death was not considered to be an SAE, but the result of one. Failure to achieve return of spontaneous circulation was not considered to be an SAE. Additional events that did not qualify for reporting as SAEs were re-arrests occurring within 24 hours and deaths directly due to lack of cardiac or neurological recovery from the index event.
Arm/Group | RhinoChill | Control
Serious Adverse Events (participants affected / at risk) | 6 | 12
Other Adverse Events (participants affected / at risk) | 17/96 | 3/104
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | RhinoChill | Control
Acute Myocardial Infarct (Cardiac disorders) | 2/27 (2) | 1/32 (1) — new; occurring more than 24 hours after hospitalization
Bleeding (Blood and lymphatic system disorders) | 1/96 (1) | 1/104 (1) — Bleeding could occur from any orifice
Convulsions (Nervous system disorders) | 1/96 (1) | 1/104 (1)
Lethal/long-lasting arrhythmia (Cardiac disorders) | 1/27 (1) | 2/32 (2)
Metabolic acidosis (General disorders) | 0/27 (0) | 2/32 (2)
Renal Failure (Renal and urinary disorders) | 1/27 (1) | 2/32 (2)
Sepsis/Multi-organ failure (General disorders) | 0/27 (0) | 3/32 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | RhinoChill (N=96) | Control (N=104)
Arrhythmia (Cardiac disorders) | 0/27 (0) | 1/32 (1)
Bleeding (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Nasal discoloration (Skin and subcutaneous tissue disorders) | 13 (13) | 0 (0)
Peri-orbital emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less